CLINICAL TRIAL: NCT03173872
Title: The Acceptance of Reiki Therapy as a Complementary and Alternative Option for the Management of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr MeLisa Gantt, LTC (Ret.) MeLisa Gantt, Landstuhl Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-10617
Record Dates: First submitted 2017-04-17; First posted 2017-06-02 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Pain, Chronic
Keywords: Reiki; Chronic Pain; Military
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: A short prospective, exploratory one group study to assess the acceptance of Reiki in 30 military healthcare beneficiaries, by comparing pre and post Reiki intervention measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One Group Study Arm (Experimental): One group study arm assesses pre Reiki and post Reiki intervention measures
  Interventions: Procedure: Reiki Protocol Hand Placement Procedures

INTERVENTIONS:
Procedure: Reiki Protocol Hand Placement Procedures — Ten Reiki hand placement procedures will last 3 minutes each for a total Reiki session lasting 30 minutes long.

SUMMARY:
For the past few years, the military has been looking for an innovative way to decrease the use of opioids for chronic pain. This has prompted military treatment facilities to begin integrating complementary and/or alternative medicine modalities into their conventional plans of care. Reiki, a bio-field energy therapy, is one such modality. The purpose of this prospective repeated measure study is to: 1) introduce the concept Reiki therapy to military healthcare beneficiaries experiencing chronic pain, 2) assess pain outcome after receiving six treatments of Reiki therapy, and 3) assess participant's impression of Reiki therapy as a possible complementary and/or alternative option for the management of chronic pain.

Thirty military healthcare beneficiaries with the complaint of chronic pain will receive a brief introduction to Reiki therapy followed by six 30-minute Reiki sessions provided by trained Reiki Level 1 Practitioner. Participant's knowledge of Reiki will be assessed using pre and post questionnaires; pain will be assessed using the Brief Pain Inventory, Defense Veterans Pain Rating Scale, DoD (Department of Defense) VA (Veteran's Administration) Pain Supplementary Questionnaire, McGill Pain Questionnaire and pain medication diaries; and participant's impression will be assessed using the Patient Global Impression of Improvement Scale and along with a post study questionnaire. If it is found that Reiki therapy helped in decreasing chronic pain outcomes, this treatment modality may be added to Landstuhl Regional Medical (LRMC) Pain Clinic's pool of complementary and alternative medicine options.

ELIGIBILITY:
Inclusion Criteria:

1. Has chronic pain (defined as pain that lasts 3 months or more since first onset).
2. Is receiving a stable pain medication regimen (defined as a regimen that has not increased 10% to 20% in the past week prior to enrollment), if on pain medication.
3. Is affiliated with at least one of the 13 installations within the Kaiserslautern Military Community area
4. Is eligible to receive healthcare at Landstuhl Regional Medical Center
5. Is 18 years and older
6. Can read and speak English
7. Is able to commit to 6 treatments (approximately 2-3 weeks)

Exclusion Criteria:

1. Have had surgery or a painful procedure in the last 30 days or are being scheduled for any surgeries or painful procedures during the duration of the study
2. Already have a working knowledge (e.g., credentialed Reiki Level I, II or III Practitioner or Reiki Master) of Reiki or have had Reiki therapy in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Pain Description, Relief and Interference with Daily Life (via Brief Pain Inventory) | From baseline measure to up to 3 weeks
  This instrument assesses the time relation sensory component of pain intensity (average over the last week, worst and least, and present pain) using a numeric rating scale (0 [No pain] to 10 [Pain as bad as you can imagine]), percentage of pain relief (0 [No relief] to 100% [Complete relief]), and 7 pain interferences concerning work, activity, mood, enjoyment, sleep, walk and relationships are assessed using 0-10 numeric scales (0 [No interference] to 10 [Complete interference]).

SECONDARY OUTCOMES:
Sensory and Affective Pain Perception (via McGill Pain Questionnaire) | From baseline measure to up to 3 weeks
  This instrument is a brief screening tool for pain and has 3 subscales: Sensory (11 word items), Affective (4 word items), and a composite Evaluative score. Fifteen words represent acute, intermittent and chronic pains, and are scored on a four-point Likert-type scale from 0 = none to 3 = severe. A total score of 45 is possible by summing the Sensory and Affective subscales and scoring them separately.
Current Pain Level (Defense and Veteran Pain Rating Scale) | From baseline measure to up to 3 weeks
  A Likert Scale graphic tool to describe one's "current" level of pain. The score ranges from 0 "no pain" to 10 "as bad as it could be nothing else matter". The scale is also colored coated depicting Mild 1-3 (Green), Moderate 4-7 (Yellow) and Severe 8-10 (Red).
Impression of current pain's affect on sleep, mood and stress (via DoD/VA Pain Supplemental Questionnaire) | From baseline measure to up to 3 weeks
  This 4-item Likert Scale instrument is used in conjunction with the Defense and Veteran Pain Rating Scale to measure the biopsychosocial impact of "current" pain level on four areas… activity sleep mood and stress.
Impression of Improvement (via Patient Global Impression of Improvement Scale Questionnaire) Patient Global Impression of Improvement Scale | At mid-point measure and again at 3 weeks
  This instrument consists of a 7-point Likert scale with 1 = "very much improved" to 7 = "very much worse" to capture overall changes related to a study medication or intervention.
Knowledge About Reiki (via Reiki Knowledge Assessment Questionnaire) | From baseline measure to up to 3 weeks
  This 5-item questionnaire to measure the participant's knowledge about Reiki. The instrument asks five of the most commonly missed questions regarding Reiki…the definition, history, credentials of practitioner, origin and usage.
Willingness to inform other about Reiki and to continue treatments (via Reiki Post Study Questionnaire) | At the conclusion of 3 weeks
  This 5-item questionnaire assesses the participant's impression of Reiki, their willingness to tell a family member, friend or co-worker about the therapy; and their thought of Reiki being offered a permanent treatment option at their healthcare facility.

CONTACTS AND LOCATIONS:
Overall Officials: MeLisa A Gantt, PhD, Principal Investigator — Gantt Clinical Research Institute LLC
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Germany

IPD SHARING:
Plan to Share IPD: Undecided